CLINICAL TRIAL: NCT06007118
Title: Adjuvant Partial-breast Irradiation of Early-stage Breast Cancer Using Stereotactic Body Radiation Therapy
Brief Title: Adjuvant Partial-breast Irradiation Using Stereotactic Body Radiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masaryk Memorial Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NV19-03-00354
Record Dates: First submitted 2023-07-20; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-07

CONDITIONS: Early-stage Breast Cancer
Keywords: breast cancer; adjuvant radiotherapy; accelerated partial breast irradiation; surgical bed
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The trial is designed as binary outcome parallel group non-inferiority trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APBI, accelerated partial breast irradiation (Experimental): The APBI group will be irradiated with a dose of 30Gy in 5 fractions in 5 working days.
  Interventions: Radiation: APBI
- WBI, whole breast irradiation (Active Comparator): The control group of patients will be irradiated with a standard accelerated mode within 20 working days.
  Interventions: Radiation: WBI

INTERVENTIONS:
Radiation: APBI — accelerated partial breast irradiation to the surgery bed (5 x 6,0 Gy; in 5 working days)
  Arms: APBI, accelerated partial breast irradiation
Radiation: WBI — accelerated whole breast irradiation with the boost to tumor bed (15x 2,67 Gy + 5x 2,0 Gy, every working day)
  Arms: WBI, whole breast irradiation

SUMMARY:
The adjuvant radiotherapy (RT) of the early-stage breast cancer patients as local treatment aims to eliminate the potential microscopic residual disease in the surgery bed or satellites in its neighborhood. Nowadays accelerated partial breast irradiation (APBI) is recommended for highly selected patients. This prospective randomized study compares the targeted external beam APBI with commonly used accelerated whole-breast irradiation (WBI) in terms of feasibility, safety, tolerance, and cosmetic effects. It is designed as non-inferiority trial and its aim is to increase the level of evidence for establishment of external beam APBI in indicated patients into daily clinical practice.

DETAILED DESCRIPTION:
Early-stage breast cancer patients after partial mastectomy are screened for eligibility. The inclusion criteria are age ˃ 50 years, non-lobular carcinoma histology, size ≤ 2 cm, negative margins ≥ 2 mm, L0, ER-positive, HER-2 negative. Enrolled patients are equally randomized into two arms according to radiotherapeutic regiment - external beam APBI (5× 6 Gy) and accelerated whole breast irradiation with the boost (15× 2,67Gy + 5× 2Gy). The follow-up visits are planned at the end of RT and 1, 3, 6, 9, and 12 months after radiation, in the second year every 4 months and then every 6 months. Cosmetics results and toxicity are evaluated using questionnaires, CTCAE criteria, and photodocumentation of the irradiated chest. The main objective of presented study is to evaluate the feasibility, safety, tolerance, and cosmetic effects of SBRT irradiation to the surgery bed in five fractions. In addition to standard clinical examination and evaluation of acute and late side effects, patients together with clinicians and nurses will independently complete a questionnaire on the impact of irradiation on the cosmetic effect. The technique of targeted external beam APBI should demonstrate better feasibility and less toxicity than the standard regimen in the adjuvant setting in treating early-stage breast cancer patients. Consequently, the presented study should increase the level of evidence for RT-indicated patients to the establishment of external APBI into daily clinical practice.

ELIGIBILITY:
Patients referred to medical attention for adjuvant radiotherapy of early-stage breast cancer at the Department of Radiation Oncology, Masaryk Memorial Cancer Institute (MMCI) were screened for eligibility. If all inclusion/exclusion criteria will be met, they were invited to participate in the present study.

Inclusion Criteria:

1. Age ≥50 years
2. Karnofsky index > 70
3. Partial mastectomy (breast-conserving surgery)
4. DCIS G1/2 ≤ 2.5 cm with negative margins (≥ 3 mm) or invasive (non-lobular) luminal-like HER2 negative carcinoma ≤ 2 cm with negative margins (≥ 2 mm) without LVI
5. In the case of invasive carcinoma, performing of axillary dissection (≥6 negative lymph nodes) or negative sentinel node biopsy

Exclusion Criteria:

1. Prior to other chest or breast surgery (including breast reconstruction), the absence of surgical clips in the tumor bed
2. Prior ipsilateral chest or breast radiotherapy
3. Neoadjuvant systemic therapy
4. Adjuvant chemotherapy
5. Multifocal or multicentric involvement
6. BRCA 1 or 2 mutations or known mutations in other high penetrance genes
7. Any systemic illness (collagen vascular diseases) or unstable medical condition that might pose additional risks for the performance of radiotherapy including claustrophobia or jactation
8. Any other factors that, in the opinion of the site investigators, would interfere with adherence to study requirements
9. Pregnancy or breastfeeding
10. Inability or unwillingness of the subject to sign written informed consent

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
APBI vs. WBI - toxicity | 44 months
  Comparison of acute and late toxicity of the APBI of the early stage breast cancer with accelerated irradiation regimen.
APBI vs. WBI - cosmetic effects | 44 months
  Comparison of cosmetic effects of the APBI of the early stage breast cancer with accelerated irradiation regimen. Cosmetic effects independently evaluated by patient, physician, and nurse scored using Harvard scale (4-point Likert scale). The scale contains 4 values - nearly identical as untreated (the best outcome), slightly different, clearly different, seriously distorted (the worst outcome)
APBI - feasibility | 44 months
  Evaluation of feasibility of the APBI regimen based on the proportion of patients who completed radiation in a total of 10 days and the proportion of patients who were irradiated exactly according to technical guidelines.
APBI vs. WBI - tolerance | 44 months
  Comparison of tolerance of the APBI of the early stage breast cancer with accelerated irradiation regimen. The toxicity was evaluated by CTCAE criteria (Common Terminology Criteria for Adverse Events). The outcome to define the tolerance a safety was CTCAE grade II or greater skin toxicity.
APBI vs. WBI - safety | 44 months
  Comparison of safety of the APBI of the early stage breast cancer with accelerated irradiation regimen. The toxicity was evaluated by CTCAE criteria (Common Terminology Criteria for Adverse Events). The outcome to define the tolerance a safety was CTCAE grade II or greater skin toxicity.

SECONDARY OUTCOMES:
Quality of life C30 | 44 months
  Quality of Life assessment using the standardized European Organisation for Research and Treatment of Cancer (EORTC) questionnaire QLQ-C30. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Quality of life BR45 | 44 months
  Quality of Life assessment using the standardized European Organisation for Research and Treatment of Cancer (EORTC) questionnaire with special module for patients with breast cancer (Breast QLQ-BR45). All of the scales and single item measures range in score from 0 to 100. A high score for the functional scales and functional single items represents a high/healthy level of functioning, whereas a high score for the symptom scales and symptom item represents a high level of symptomatology or problems.
Effectivity | 44 months
  Assessment of effectivity of the treatment method by evaluating subsequent endpoints such as LC (local control) and OS (overall survival). Overall survival (OS) is defined as the time from randomization to death from any cause. Local control (LC) is defined as the time from randomization to the first local recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Burkon, M.D., Ph.D., Principal Investigator — Masaryk Memorial Cancer Institute, Dept. of Radiation Oncology,
Locations (1):
- Masaryk Memorial Cancer Institute, Brno, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strnad V, Polgar C, Ott OJ, Hildebrandt G, Kauer-Dorner D, Knauerhase H, Major T, Lyczek J, Guinot JL, Gutierrez Miguelez C, Slampa P, Allgauer M, Lossl K, Polat B, Fietkau R, Schlamann A, Resch A, Kulik A, Arribas L, Niehoff P, Guedea F, Dunst J, Gall C, Uter W; Groupe Europeen de Curietherapie and European Society for Radiotherapy and Oncology. Accelerated partial breast irradiation using sole interstitial multicatheter brachytherapy compared with whole-breast irradiation with boost for early breast cancer: 10-year results of a GEC-ESTRO randomised, phase 3, non-inferiority trial. Lancet Oncol. 2023 Mar;24(3):262-272. doi: 10.1016/S1470-2045(23)00018-9. Epub 2023 Feb 1. PMID 36738756
- [Background] Meattini I, Marrazzo L, Saieva C, Desideri I, Scotti V, Simontacchi G, Bonomo P, Greto D, Mangoni M, Scoccianti S, Lucidi S, Paoletti L, Fambrini M, Bernini M, Sanchez L, Orzalesi L, Nori J, Bianchi S, Pallotta S, Livi L. Accelerated Partial-Breast Irradiation Compared With Whole-Breast Irradiation for Early Breast Cancer: Long-Term Results of the Randomized Phase III APBI-IMRT-Florence Trial. J Clin Oncol. 2020 Dec 10;38(35):4175-4183. doi: 10.1200/JCO.20.00650. Epub 2020 Aug 24. PMID 32840419
- [Background] Meattini I, Becherini C, Boersma L, Kaidar-Person O, Marta GN, Montero A, Offersen BV, Aznar MC, Belka C, Brunt AM, Dicuonzo S, Franco P, Krause M, MacKenzie M, Marinko T, Marrazzo L, Ratosa I, Scholten A, Senkus E, Stobart H, Poortmans P, Coles CE. European Society for Radiotherapy and Oncology Advisory Committee in Radiation Oncology Practice consensus recommendations on patient selection and dose and fractionation for external beam radiotherapy in early breast cancer. Lancet Oncol. 2022 Jan;23(1):e21-e31. doi: 10.1016/S1470-2045(21)00539-8. PMID 34973228
- [Background] Thomsen MS, Alsner J, Nielsen HM, Jakobsen EH, Nielsen MH, Moller M, Pedersen AN, Yates E, Berg M, Lorenzen E, Jensen I, Josipovic M, Overgaard J, Offersen BV; DBCG RT Committee. Volume matters: Breast induration is associated with irradiated breast volume in the Danish Breast Cancer Group phase III randomized Partial Breast Irradiation trial. Radiother Oncol. 2022 Dec;177:231-235. doi: 10.1016/j.radonc.2022.09.024. Epub 2022 Oct 17. PMID 36265685
- [Background] Vicini FA, Cecchini RS, White JR, Arthur DW, Julian TB, Rabinovitch RA, Kuske RR, Ganz PA, Parda DS, Scheier MF, Winter KA, Paik S, Kuerer HM, Vallow LA, Pierce LJ, Mamounas EP, McCormick B, Costantino JP, Bear HD, Germain I, Gustafson G, Grossheim L, Petersen IA, Hudes RS, Curran WJ Jr, Bryant JL, Wolmark N. Long-term primary results of accelerated partial breast irradiation after breast-conserving surgery for early-stage breast cancer: a randomised, phase 3, equivalence trial. Lancet. 2019 Dec 14;394(10215):2155-2164. doi: 10.1016/S0140-6736(19)32514-0. Epub 2019 Dec 5. PMID 31813636
- [Background] Olivotto IA, Whelan TJ, Parpia S, Kim DH, Berrang T, Truong PT, Kong I, Cochrane B, Nichol A, Roy I, Germain I, Akra M, Reed M, Fyles A, Trotter T, Perera F, Beckham W, Levine MN, Julian JA. Interim cosmetic and toxicity results from RAPID: a randomized trial of accelerated partial breast irradiation using three-dimensional conformal external beam radiation therapy. J Clin Oncol. 2013 Nov 10;31(32):4038-45. doi: 10.1200/JCO.2013.50.5511. Epub 2013 Jul 8. PMID 23835717
- [Background] Murray Brunt A, Haviland JS, Wheatley DA, Sydenham MA, Alhasso A, Bloomfield DJ, Chan C, Churn M, Cleator S, Coles CE, Goodman A, Harnett A, Hopwood P, Kirby AM, Kirwan CC, Morris C, Nabi Z, Sawyer E, Somaiah N, Stones L, Syndikus I, Bliss JM, Yarnold JR; FAST-Forward Trial Management Group. Hypofractionated breast radiotherapy for 1 week versus 3 weeks (FAST-Forward): 5-year efficacy and late normal tissue effects results from a multicentre, non-inferiority, randomised, phase 3 trial. Lancet. 2020 May 23;395(10237):1613-1626. doi: 10.1016/S0140-6736(20)30932-6. Epub 2020 Apr 28. PMID 32580883
- [Background] Whelan TJ, Julian JA, Berrang TS, Kim DH, Germain I, Nichol AM, Akra M, Lavertu S, Germain F, Fyles A, Trotter T, Perera FE, Balkwill S, Chafe S, McGowan T, Muanza T, Beckham WA, Chua BH, Gu CS, Levine MN, Olivotto IA; RAPID Trial Investigators. External beam accelerated partial breast irradiation versus whole breast irradiation after breast conserving surgery in women with ductal carcinoma in situ and node-negative breast cancer (RAPID): a randomised controlled trial. Lancet. 2019 Dec 14;394(10215):2165-2172. doi: 10.1016/S0140-6736(19)32515-2. Epub 2019 Dec 5. PMID 31813635
- [Background] Coles CE, Griffin CL, Kirby AM, Titley J, Agrawal RK, Alhasso A, Bhattacharya IS, Brunt AM, Ciurlionis L, Chan C, Donovan EM, Emson MA, Harnett AN, Haviland JS, Hopwood P, Jefford ML, Kaggwa R, Sawyer EJ, Syndikus I, Tsang YM, Wheatley DA, Wilcox M, Yarnold JR, Bliss JM; IMPORT Trialists. Partial-breast radiotherapy after breast conservation surgery for patients with early breast cancer (UK IMPORT LOW trial): 5-year results from a multicentre, randomised, controlled, phase 3, non-inferiority trial. Lancet. 2017 Sep 9;390(10099):1048-1060. doi: 10.1016/S0140-6736(17)31145-5. Epub 2017 Aug 2. PMID 28779963
- [Background] Meattini I, Poortmans PMP, Marrazzo L, Desideri I, Brain E, Hamaker M, Lambertini M, Miccinesi G, Russell N, Saieva C, Strnad V, Visani L, Kaidar-Person O, Livi L. Exclusive endocrine therapy or partial breast irradiation for women aged >/=70 years with luminal A-like early stage breast cancer (NCT04134598 - EUROPA): Proof of concept of a randomized controlled trial comparing health related quality of life by patient reported outcome measures. J Geriatr Oncol. 2021 Mar;12(2):182-189. doi: 10.1016/j.jgo.2020.07.013. Epub 2020 Jul 29. PMID 32739355
- [Derived] Burkon P, Selingerova I, Vrzal M, Holanek M, Coufal O, Polachova K, Andraskova V, Jhawar SR, Slampa P, Kazda T, Slavik M. Quality of life in early breast cancer patients after adjuvant accelerated partial-breast irradiation (APBI) in randomized trial. Sci Rep. 2025 Jan 9;15(1):1387. doi: 10.1038/s41598-025-85342-2. PMID 39779797
- [Derived] Burkon P, Selingerova I, Slavik M, Holanek M, Vrzal M, Coufal O, Polachova K, Muller P, Slampa P, Kazda T. Toxicity of external beam accelerated partial-breast irradiation (APBI) in adjuvant therapy of early-stage breast cancer: prospective randomized study. Radiat Oncol. 2024 Feb 3;19(1):17. doi: 10.1186/s13014-024-02412-x. PMID 38310249